CLINICAL TRIAL: NCT04154410
Title: Prospective Observational Study of the Non Invasive Objective Assessment of Pre-operative Anxiety Using the Heart Rate Variability and the Pupillary Reflex Measurement
Brief Title: Prediction of Pre-operative Anxiety by Heart Variability and Pupillometry
Acronym: INNOVANX
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190697; 2019-A01743-54 (Other: ID-RCB)
Record Dates: First submitted 2019-09-23; First posted 2019-11-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Eligible for Day Case Surgery
Keywords: Pre-operative anxiety; pupillometry; heart rate variability; cardiac coherence state; ambulatory surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Analgesia Nociception Index — Non invasive finger tip monitoring before during and 5 minutes after cannulation
  Other Names: Heart rate variability measures
Other: algiscan — Portable videopupillometer to measure pupillary light reflex (PLR), variation coefficient of pupillary diameter (VCPD), pupillary diameter (PD) fluctuations before, during and 5 minutes after cannulation
  Other Names: Pupillometric measures

SUMMARY:
The purpose of this study is to determine whether heart rate variability levels and pupillometric measures are effective objective predictors of anxiety among patients before surgery.

DETAILED DESCRIPTION:
The prevalence of preoperative anxiety in adults is estimated between 60 and 80% and prevents a good integration of the information delivered, while seeking more attention from caregivers. In addition, anxious patients require the administration of higher doses of hypnotics at anesthetic induction. The pain expressed in the postoperative period is proportional to preoperative anxiety, with a slower recovery kinetics responsible for prolonged stay in the recovery room. Finally, the incidence of chronic pain is correlated with the intensity of preoperative anxiety.

While the recommendations of the European Anesthesia Society (ESA) emphasize the importance of managing preoperative anxiety, this dimension is often overlooked and existing methods of assessment are time consuming and sometime inaccurate.

Objective screening with dynamic monitoring of the level of anxiety in real time is the necessary step to ensure accurate detection and personalized management of the emotional state of patients before performing an invasive procedure.

Anxiety is an emotional state reflecting an imbalance of cortico-frontal regulation on the limbic system. The interaction between these two neuronal systems is expressed in particular by the intensity of the vagal tone and the autonomic nervous system. Exploring the balance between sympathetic and parasympathetic systems is a promising avenue of exploration for identifying, predicting, and treating anxiety.

Two reliable and easy-to-use devices analyzing the expression of the autonomic nervous system validated in the analysis of nociception in the awake patient or under general anesthesia are marketed:

A. Analgesia Nociception Index (ANI) (MDoloris Medical Systems) analyzing oscillatory changes in heart rate as a function of respiratory time, namely the heart rate variability (HRV) B. Algiscan (IDMed) analyzing pupil responsiveness to nociception

The use of these devices in conscious pre-operative patients could allow a reliable and objective detection of anxiety while following its kinetic evolution over time. The purpose of this project is to evaluate the validity of these two devices in the context of preoperative anxiety. After receiving clear information and giving their written agreement, patients will be included in the study by the anesthetist physician. During the anesthesia consultation, the included patients will be subjected to a Surgical Fear Questionnaire (SFQ) questionnaire of level of anxiety.

A secondary study will consist of connecting a lighting device connected to the heart rate variability to emit a relaxing light in the preoperative waiting room.

ELIGIBILITY:
Inclusion Criteria:

-Day case surgical patients

Exclusion Criteria:

* <18yo
* psychiatric disorders
* participating refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective patients for day-case surgical procedure
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Analgesia Nociception Index (ANI) | at Day 0
  Index from 0 to 100 Variation 5 minutes before during and 5 minutes after cannulation Comparison between anxious and non-anxious patients Measure of anxiety reduction

SECONDARY OUTCOMES:
Coefficient of variation of pupillary diameter (CVDP) | at Day 0
  Percentage from 0 to 100% Variation 5 minutes before during and 5 minutes after cannulation Comparison between anxious and non-anxious patients
Visual Analog Scale (VAS) | at Day 0
  Measure of anxiety reduction 30 minutes after the beginnig of the luminous immersion
Heart rate variability | at Day 0
  comparison between anxious and non-anxious patients Variation 5 minutes before during and 5 minutes after cannulation
Analgesia Nociception Index (ANI) | at Day 0 - after 30 minutes immersive light intervention
  Impact of 30 minutes immersive light intervention on measures of ANI and VAE
Visual Analog Scale (VAS) | at Day 0 - after 30 minutes immersive light intervention
  Impact of 30 minutes immersive light intervention on measures of ANI and VAS

CONTACTS AND LOCATIONS:
Overall Officials: Gilles GUERRIER, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cochin Hospital, APHP, Paris, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richez J, Rothschild PR, Baillard C, Guerrier G. Investigating pupillometry to detect preoperative anxiety: a pilot study. Front Psychol. 2024 Jan 3;14:1296387. doi: 10.3389/fpsyg.2023.1296387. eCollection 2023. PMID 38239470